CLINICAL TRIAL: NCT02628704
Title: Phase 2, Randomized, Double-blind, Placebo-controlled, Multicenter Study of Selinexor (KPT-330), Carfilzomib, and Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma Previously Treated With a Proteasome Inhibitor and an Immunomodulatory Drug
Brief Title: Selinexor, Carfilzomib, and Dexamethasone Versus Placebo, Carfilzomib, and Dexamethasone in Multiple Myeloma
Acronym: SCORE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KCP-330-015
Record Dates: First submitted 2015-12-02; First posted 2015-12-11 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma
Keywords: Karyopharm; selinexor; KPT-330; multiple myeloma; SCORE
MeSH Terms: conditions — Multiple Myeloma | interventions — selinexor; carfilzomib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selinexor, carfilzomib and dexamethasone (Experimental): 60 mg of selinexor and and 20 mg of dexamethasone will be taken twice weekly. On days coinciding with carfilzomib administration, selinexor will be given between 30 minutes and 4 hours after the end of the carfilzomib infusion.
  Interventions: Drug: Selinexor; Drug: carfilzomib; Drug: Dexamethasone
- Placebo, carfilzomib and dexamethasone (Placebo Comparator): Placebo (for 60 mg of selinexor) and and 20 mg of dexamethasone will be taken twice weekly. On days coinciding with carfilzomib administration, Placebo (for 60 mg of selinexor) will be given between 30 minutes and 4 hours after the end of the carfilzomib infusion.
  Interventions: Drug: Placebo (for selinexor); Drug: carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Selinexor — The fixed dose of selinexor is 60 mg (three 20 mg tablets)
  Other Names: KCP-330
  Arms: Selinexor, carfilzomib and dexamethasone
Drug: Placebo (for selinexor) — sugar tablet manufactured to mimic selinexor tablet
  Arms: Placebo, carfilzomib and dexamethasone
Drug: carfilzomib — Administered as an IV infusion on Days 1, 2, 8, 9, 15 and 16 of each 4-week cycle for Cycles 1-13 and then on Days 1, 2, 15, and 16 for Cycles ≥ 14.
  Other Names: Kyprolis
Drug: Dexamethasone — Fixed oral dose of 20 mg will be given twice weekly (Days 1, 2, 8, 9, 15, 16, 22 and 23) in each cycle.

SUMMARY:
Double-blind study will compare the efficacy and assess safety of selinexor plus carfilzomib (Kyprolis®) plus low-dose dexamethasone versus placebo plus carfilzomib plus low-dose dexamethasone in patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a Phase 2, two-arm, randomized, placebo-controlled, double-blind, multicenter study of relapsed/refractory multiple myeloma patients who have received at least two prior therapies, including a proteasome inhibitor and an IMiD.

Patients who meet all the eligibility criteria will be randomized to one of two blinded treatment arms:

* selinexor + carfilzomib + dexamethasone
* placebo + carfilzomib + dexamethasone

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, histologically confirmed MM, based on IMWG guidelines. Patients must have measurable disease as defined by at least one of the following:

  * Serum M-protein ≥ 1.0 g/dL by serum protein electrophoresis (SPEP) or for immunoglobulin (Ig) A myeloma, by quantitative IgA; or
  * Urinary M-protein excretion at least 200 mg/24 hours; or
  * Serum FLC ≥ 100 mg/L, provided that the serum FLC ratio is abnormal.
  * If serum protein electrophoresis is felt to be unreliable for routine M- protein measurement, then quantitative Ig levels by nephelometry or turbidometry are acceptable.
* Must have received ≥ 2 prior anti-MM therapies including a proteasome inhibitor and an IMiD. The most recent proteasome inhibitor must not have been carfilzomib.
* Patients previously treated with carfilzomib are eligible as long as they meet the following criteria:

  * Not received carfilzomib within 6 months (183 days) of Cycle 1 Day 1 (C1D1), and
  * Carfilzomib was not part of their most recent therapy for the treatment of MM, and
  * Did not discontinue carfilzomib treatment because of adverse effects.
* MM that is refractory to the most recent treatment regimen. Refractory is defined as ≤ 25% response to therapy, or progression during therapy, or progression on or within 60 days after completion of therapy.

Exclusion Criteria:

* Smoldering MM.
* Active plasma cell leukemia.
* MM that does not express M-protein or serum FLC (i.e., non-secretory MM is excluded; plasmacytomas without M-protein or serum FLC are excluded).
* Documented active systemic amyloid light chain amyloidosis.
* Active MM involving the central nervous system.
* Active polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome.
* Prior autologous stem cell transplantation < 1 month or allogenic stem cell transplantation < 3 months prior to C1D1.
* Active graft versus host disease (after allogeneic stem cell transplantation) at C1D1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Assessed from the date of first dose of blinded study treatment until the date that PD assessed up to 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - James R. Berenson MD, Inc, West Hollywood, California
  - Waverly Hematology, Cary, North Carolina

IPD SHARING:
Plan to Share IPD: Yes